CLINICAL TRIAL: NCT02351570
Title: Offer and Mediation of §20 SGB V Health Prevention Programmes to Patients Through Their Treating General Practitioner - a Mixed Methods Study
Brief Title: Health Prevention Programmes to Patients Through Their General Practitioners
Status: Completed | Type: Observational
Sponsor: Berlin School of Public Health (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christine Holmberg, Dr phil, Berlin School of Public Health
Other Study IDs: BSPH GP´s Prevention Programme
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Prevention

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
By the health reform GKV in 2000 as well as by the competitive strengthening law GKV in 2007 in §20 SGB V the health insurance schemes have received an enlarged action frame in the primary prevention and the operational health support.

Through these paragraphs arises the possibility for citizens to let refund health-supporting programmes or health training of the health insurance schemes.

Doctor's recommendation is one of the most important predictors by therapy decisions of patients.

At the same time, primary prevention takes a very small part of the working hours of general practitioners.

Hence, is the aim of the present study to examine whether and how general practitioners could be incorporated in the mediation of prevention's offers.

To reach this aim, must be grasped first, to what extent general practitioners are already integrated into in the mediation of the primary prevention courses. There is up to now no information about whether general practitioners know about the GKV-improved prevention programmes for GKV-insured person and whether they are involved in their mediation. This research project will close this gap.

The aims of the study are:

1. to explore the roll of primary prevention in the general practitioner's consultation
2. to analyse which social institutions are responsible for primary prevention according to the general practitioner's opinion
3. to explore which primary prevention's programmes do general practitioners in their consultation recommend
4. to analyse which factors play a role in the mediation
5. to explore whether general practitioners with §20 are familiar.

This is a mixed methods study which combines a mail survey of all general practitioners in Berlin with focus groups of 25 general practitioners.

In this study all general practitioners of Berlin (n=1300) will be mailed. Participants for the focus groups are invited from the pool of teaching doctors of the Institute for General Medicine at the Charite.

After both methods are analyzed on their own, the triangulation of the interpretation of both data sets will be done to find possible answers of the study questions. Bi-directionality of results will contribute to find possible interpretations of the survey responses in the results of the focus group discussions, as well as the results of the focus groups discussions could be explained by the results of the survey (Flick).

DETAILED DESCRIPTION:
Background In Germany 70% of the men and 50% of the women are overweight or obese. On account of the frequency of overweight, diabetes and other life style-related risk factors and the raised risk linked with it for chronic illnesses it has been initiated preventive measures.

By the health reform GKV in 2000 as well as by the competitive strengthening law GKV in 2007 in §20 SGB V the health insurance schemes have received an enlarged action frame in the primary prevention and the operational health support.

Through these paragraphs arises the possibility for citizens to let refund health-supporting programmes or health training of the health insurance schemes. Moreover programmes count to the support of physical activity, nutrition consultation, smoke weaning programmes or also learning of relaxation techniques. About two to three percent of all GKV insured person take part in primary-preventive courses and seminar offers.

Doctor's recommendation is one of the most important predictors by therapy decisions of patients.

At the same time, primary prevention takes a very small part of the working hours of general practitioners.

Hence, is the aim of the present study to examine whether and how general practitioners could be incorporated in the mediation of prevention's offers.

To reach this aim, must be grasped first, to what extent general practitioners are already integrated into in the mediation of the primary prevention courses. There is up to now no information about whether general practitioners know about the GKV-improved prevention programmes for GKV-insured person and whether they are involved in their mediation. This research project will close this gap.

The aims of the study are:

1. to explore the roll of primary prevention in the general practitioner's consultation
2. to analyse which social institutions are responsible for primary prevention according to the general practitioner's opinion
3. to explore which primary prevention's programmes do general practitioners in their consultation recommend
4. to analyse which factors play a role in the mediation
5. to explore whether general practitioners with §20 are familiar.

Methods

1. Study design:

   This is a mixed methods study which combines a mail survey of all general practitioners in Berlin with focus groups of 25 general practitioners.

   The design arises from the study question, so that we grasp from the mail survey to what extent primary prevention in the general practitioner's practice a role plays and whether §20 is known among general practitioners.

   In the focus groups will be analyzed which role can or want general practitioners in the primary prevention take and to what extent they can perceive themselves as mediators with regard to the offer of §20 programms. Barriers as well as the role of the general practitioner in the primary prevention will be explored.
2. Study population In this study all general practitioners of Berlin (n=1300) will be mailed. Participants for the focus groups are invited from the pool of teaching doctors of the Institute for General Medicine at the Charite (see characteristics below) which are also part of the mail survey.

   Characteristics of teaching doctors of the general medicine Charité Berlin:
   * Aptitude and joy in teaching
   * Specialist in general medicine, general practice internist or active internist
   * Duration of establishment > 3 years
   * More than 500 GKV-Versicherte / quarter
   * Typical general practitioner spectrum without one-sided practice
   * Regular house visits
   * Separate space for students
   * Guarantee of the necessary number of hours
3. Procedure Survey For the data collection a standardized questionnaire was developed. A literature research as well as the objective of the study led the questionnaire development. After its completion the comprehensibility of the questionnaire was checked with cognitive interviews.

   Data collection All 1300 general practitioners in Berlin are written up by the service provider Data-B through the Berlin medical association.

   General practitioners will receive the validated questionnaire, a franked envelope and a franked postcard. The survey is conceived pseudonym. There will be no possibility to connect the questionnaire with personal data.

   The response rate by physician's survey rises if the survey is supported by professional associations or other prominent representatives of the field. Hence, the survey is supported by Professor Braun the Director of the Institute of General Medicine at the Charite Medical University in Berlin.

   Also the length of the questionnaire has influence on the response rate. This was considered in the development of the questionnaire.

   To raise further the response rate, we will apply the Dillman Method. This meant that we will send after three weeks a postcard reminder to the non-responders. Other two weeks later, we will send again, to those who have not answered, the questionnaire as well as the franked postcard. Those general practitioners that after 4 weeks haven't sent the postcard will be considered as non-responders.

   The franked postcard is to have an overview of which doctors have responded to the questionnaire. An identification number on the postcard allows the service provider Data-B to identify the doctor's address or practice.

   We collect for the service provider the identification number of the postcards. Data-B will send within two weeks a reminder to those whose number is not on the list.

   This procedure is carried out after two weeks once again, but this time with the questionnaire. Because this is the third and last contact, no postcard is included in this last mailing.

   The data of the questionnaire are administered by the BSPH and the address file by Data-B. With it is the pseundonymity of the survey guaranteed. For the BSPH is not possible to identify which physician has responded to which questionnaire.

   The study-staff will enter the date of the questionnaires in an Access data bank. To carry out the data analysis, the data bank will be then export to SPSS.

   Focus Groups In addition, five focus groups with five participants will be carried out. The focus groups are so structured that the different practice forms, group practice, practice with additional offers or practice with private patients are enclosed in the focus groups equally.

   So far possibly single focus groups will be composed from participants with different practice characteristic as well as age-mixed.

   Before the discussion, the participants of the focus groups are asked to fill out the questionnaire, so that it will be possible to get in contact the questionnaires with the focus groups. The questionnaires are filled and collected without personal data. Hence, it will not be possible to know which participant filled which questionnaire out.

   To be able to draw conclusion on the generalizability of the focus group's results, it will be possible to compare aggregated data of the focus groups with regard to the questionnaires with the data of the general practitioners in Berlin.

   A moderator will guide the group in the discussion and a coworker will be the observer, documenting the meeting. The focus-group process will be conducted based on a catalog of guiding questions (Annex) that will be given to the moderator at the beginning of the meeting. The Observer and the Moderator will write up a complete protocol immediately after the meeting.

   The discussions will be audio-recorded digitally. After the focus-group meeting, names and other person identifiable content will be erased from the audio-recording (by deleting or new recording) and the final audio-documents will be saved on a secure Charité Server. For each focus-group, characteristics of the practice, age structure and gender will be documented and assigned. Names of participants will not be saved.
4. Data analysis

Questionnaire A descriptive statistical analysis of the collected data will be conducted using SPSS.

Focus group discussion The content of the focus groups will be analyzed based on the catalogue of guiding questions.

The analytical procedure includes assignment of codes and application of Grounded Theory. This open process of the analysis is chosen to allow identifying topics and relationships that might not be identified with a pure content analysis.

Triangulation After both methods are analyzed on their own, the triangulation of the interpretation of both data sets will be done to find possible answers of the study questions. Bi-directionality of results will contribute to find possible interpretations of the survey responses in the results of the focus group discussions, as well as the results of the focus groups discussions could be explained by the results of the survey (Flick).

Data confidentiality For the quantitative part of the study no person data or contact information (name, birthdates, address, phone number, email) will be collected. (see previous section). Gender and categories-based age are collected. The survey is anonymous at all stages of data collection, analysis and publication. Publications will include statistical analysis of conglomerated data. Adherence to German legislation of confidentiality is granted at all times.

Informed consent The response of completed questionnaires in the quantitative part of the study is valued as the informed consent. The postal card with the stamp of the practice allows Data-B to compare these with the Databank of names and addresses of physicians. There is impossible to identify questionnaire and practice at any time. The appearance for the focus group meeting is valued as the acceptance of participation.

The questionnaires and the digital recordings of the focus groups will be kept for 10 years at the Charité.

Ethic Committee In case that the "Datenschutzbeauftragte" of the Charity requires it, the approval of the ethic committee will be obtained. In any case the Ethic Committee will be informed of the study intended.

ELIGIBILITY:
Inclusion Criteria for Focus Groups:

* Teaching doctors of the Institute for General Medicine at the Charite
* Aptitude and joy in teaching
* Specialist in general medicine, general practice internist or active internist
* Duration of establishment > 3 years
* More than 500 GKV-Versicherte / quarter
* Typical general practitioner spectrum without one-sided practice
* Regular house visits
* Separate space for students
* Guarantee of the necessary number of hours

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study all general practitioners of Berlin (n=1300) will be mailed. Participants for the focus groups are invited from the pool of teaching doctors of the Institute for General Medicine at the Charite (see characteristics below) which are also part of the mail survey.
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
prevalence and practice of primary prevention in primary care | immediatly
  cross-sectional survey at one time point

CONTACTS AND LOCATIONS:
Locations (1):
- Berlin School of Public Health, Charite Universitätsmedizin Berlin, Berlin, State of Berlin, Germany